CLINICAL TRIAL: NCT03277430
Title: Uterus Transplantation From Live Donors and From Deceased Donors - Clinical Study
Acronym: UTxLD/DBD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: University Hospital, Motol (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Jiri Fronek, MD PhD Assoc Prof, Institute for Clinical and Experimental Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2044/15 (NM-15-01)
Record Dates: First submitted 2017-09-04; First posted 2017-09-11 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Mayer Rokitansky Kuster Hauser Syndrome; Mullerian Aplasia; Uterus; Absence, Congenital; Infertility, Female; Uterus Absence, Acquired; Absolute Uterine Factor Infertility
Keywords: uterus transplantation, absolute uterine factor infertility
MeSH Terms: conditions — Mullerian aplasia; Infertility, Female | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Live donor uterus transplantation (Experimental): Transplantation of uterus from a living donor. Immunosuppression with tacrolimus.
  Interventions: Procedure: Live donor uterus transplantation; Drug: Tacrolimus
- Deceased donor uterus transplantation (Experimental): Transplantation of uterus from a deceased brain-dead donor. Immunosuppression with tacrolimus.
  Interventions: Procedure: Deceased donor uterus transplantation; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Live donor uterus transplantation — Transplantation of uterus from a living donor.
  Arms: Live donor uterus transplantation
Procedure: Deceased donor uterus transplantation — Transplantation of uterus from a deceased brain-dead donor.
  Arms: Deceased donor uterus transplantation
Drug: Tacrolimus — Maintenance immunosuppression in UTx recipient will be reduced to tacrolimus monotherapy to minimalize fetal compromise.
  Other Names: FK506

SUMMARY:
Uterus transplantation (UTx) is the only causative treatment for congenital or acquired uterus absence. Individual cases of UTx from a live donor (LD UTx) with healthy child birth performed so far showed favourable outcomes. The present study will include both LD UTx and UTx from deceased donors after brain death (DBD UTx). The aim is treatment of uterine infertility by UTx. It is is an ethically justifiable life-promoting transplantation. Twenty UTx will be performed in 2 parallel arms: 10 LD UTx and 10 DBD UTx. Immunosuppression will be administered. Phases of the UTx procedure are: in vitro fertilization - cryopreservation of embryos - uterus retrieval - UTx - follow up - embryo transfer - pregnancy - child birth - later graft hysterectomy - life long follow up. Introduction of UTx into clinical practice may enable women with uterine infertility to have their own children.

DETAILED DESCRIPTION:
Introduction: Uterus transplantation (UTx) is the only causative treatment for congenital or acquired uterus absence, i.e. absolute uterine factor infertility (AUFI). Feasibility of uterus transplantation from o live donor and possibility of healthy child birth have been proven in previous clinical study in Sweden. The present study is supposed to extend the swedish experience by including UTx from both live donors and from deceased donors after brain death.

Aim: Treatment of absolute uterine factor infertility that has no other therapy option by uterus transplantation. Extending basic knowledge on UTx. Possible introduction of UTx into clinical practice.

Indications: UTx can be offered to patients with congenital uterus absence - aplasia uteri et vaginae, also called Mullerian aplasia or Rokitansky-Mayer-Kuster-Hauser syndrome (RMKH), in whom previous neo-vagina was created. UTx can be performed also in women with acquired uterus absence on the basis of previous hysterectomy e.g. for myomas, endometriosis, post-partum bleeding, cervical cancer, uterus malformations or intrauterine adhesions. Ovarian function must be preserved and stable male partner is required for in vitro fertilization (IVF).

Ethics: Uterus retrieval from a deceased brain-dead donor does not endanger retrieval of other life-saving organs. Live donor does not loose a vitally important organ. The only alternative is adoption of a child. Surrogacy is illegal in many european countries. UTx is the only causative treatment of AUFI. It is is an ethically justifiable life-promoting transplantation. UTx improves quality of live of both the recipient and the live donor by giving an opportunity to have an own child. Board certification for this study was obtained from the Ministry of Health of the Czech Republic and from the local Ethics Committee.

Methods: Twenty UTx will be performed in total in 2 parallel arms: 10 UTx from a live donor (LD UTx) and 10 UTx from a deceased brain-dead donor (DBD UTx). Patients who have no suitable live donor will be wait-listed for a deceased donor. Compatible blood group and negative cross-match test is required. AB0 incompatible or pair exchange transplantations are also possible. Donors and recipients will be examined by clinical, laboratory and imaging methods. All diagnostic and therapeutic procedures will be performed according to a protocol. Risk and benefit will be assessed by a multi-disciplinary team. Informed consent will be signed. Time period between UTx and embryo transfer is supposed to be about 1 year depending on condition of the recipient and the graft, e.g. level of immunosuppression, rejection or infection episodes. Adverse events will be monitored and addressed. Number of possible pregnancies and child births is estimated to be up to 2. The uterus graft will be removed in the end. Overall time interval of keeping the uterus graft in situ and exposure to immunosuppressive therapy is estimated to be up to 5 years.

Immunosuppression: Induction immunosuppression is based on thymoglobuline and corticosteroids. Maintenance immunosuppression is based on tacrolimus, mycophenolate and corticosteroids. Temporary anti-infective prophylaxis will be administered. Minimalization of immunosuppression is needed before pregnancy (monotherapy with tacrolimus). Protocol cervix biopsies to look for possible rejection will be performed. Immunosuppression will be discontinued after graft hysterectomy.

Phases of the UTx procedure: in vitro fertilization (IVF phase I) - cryopreservation of embryos - uterus retrieval from a live donor or from a deceased donor - orthotopic uterus transplantation with open technique - follow up period - embryo transfer (IVF phase II) - pregnancy - child birth via Cesarian section - later graft hysterectomy - life long follow up.

Merit: Individual cases of uterus transplantation performed so far showed favourable outcomes. Introduction of UTx into clinical practice may enable women with uterine infertility to have their own children.

ELIGIBILITY:
Inclusion Criteria for UTx recipient:

* 18 - 40 years of age
* good general health
* congenital or acquired uterus absence
* desire for a child

Exclusion Criteria for UTx recipient:

* age over 40
* serious comorbidity

Inclusion Criteria for a live uterus donor:

* female
* 18 - 60 years of age
* maximum 4 child births
* maximum 1 Cesarian section
* good general health

Exclusion Criteria for a live uterus donor:

* age over 60
* hypertension with organ damage
* diabetes mellitus
* other serious comorbidity

Inclusion Criteria for a deceased brain-dead uterus donor:

* female
* age under 60
* no previous hysterectomy
* no previous uterus malignancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-10-09 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of uterus transplantation. | Until 10 live donor and 10 deceased donor uterus transplants have been performed plus approximately 5 years.
  Number of successful uterus transplantations and healthy child births. Treatment of absolute uterine factor infertility that has no other therapy option by uterus transplantation that includes in vitro fertilization and cryopreservation, uterus transplantation from a live donor or from a deceased donor, graft survival on immunosuppression, embryo transfer, pregnancy and child birth, final graft hysterectomy.

SECONDARY OUTCOMES:
Comparison of efficacy of uterus transplantation from live donors versus deceased donors. | Until 10 live donor and 10 deceased donor uterus transplants have been performed plus approximately 5 years.
  Number of successful uterus transplantations and healthy child births from live donors versus deceased donors.
Rate of adverse events after uterus transplantation | Until 10 live donor and 10 deceased donor uterus transplants have been performed plus approximately 5 years.
  Number of recipients of uterus transplantation with adverse events.
Rate of adverse events after live uterus donation | Until 10 live donor transplants have been performed plus approximately 5 years.
  Number of live donor participants after uterus retrieval with adverse events.
Rate of adverse events during pregnancy and child birth after uterus transplantation | Until 10 live donor and 10 deceased donor uterus transplants have been performed plus approximately 5 years.
  Number of children conceived and born from transplanted uterus with adverse events.
Verification of technique of uterus retrieval | Until 10 live donor and 10 deceased donor uterus transplants have been performed plus approximately 5 years.
  Verification of surgical technique of uterus retrieval from a live donor and from a deceased donor.

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Fronek, Assoc Prof, Principal Investigator — Transplant Surgery Department, Institute of Clinical and Experimental Medicine, Prague, Czech Republic
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Erman Akar M, Ozekinci M, Alper O, Demir D, Cevikol C, Meric Bilekdemir A, Daloglu A, Ongut G, Senol Y, Ozdem S, Uzun G, Luleci G, Suleymanlar G. Assessment of women who applied for the uterine transplant project as potential candidates for uterus transplantation. J Obstet Gynaecol Res. 2015 Jan;41(1):12-6. doi: 10.1111/jog.12486. Epub 2014 Sep 17. PMID 25226847
- [Background] Olausson M, Johannesson L, Brattgard D, Diaz-Garcia C, Lundmark C, Groth K, Marcickiewizc J, Enskog A, Akouri R, Tzakis A, Rogiers X, Janson PO, Brannstrom M. Ethics of uterus transplantation with live donors. Fertil Steril. 2014 Jul;102(1):40-3. doi: 10.1016/j.fertnstert.2014.03.048. Epub 2014 Apr 28. No abstract available. PMID 24784936
- [Background] Johannesson L, Dahm-Kahler P, Eklind S, Brannstrom M. The future of human uterus transplantation. Womens Health (Lond). 2014 Jul;10(4):455-67. doi: 10.2217/whe.14.22. PMID 25259905
- [Background] Farrell RM, Falcone T. Uterine transplantation. Fertil Steril. 2014 May;101(5):1244-5. doi: 10.1016/j.fertnstert.2014.03.022. Epub 2014 Apr 13. No abstract available. PMID 24726215
- [Background] Brannstrom M, Johannesson L, Dahm-Kahler P, Enskog A, Molne J, Kvarnstrom N, Diaz-Garcia C, Hanafy A, Lundmark C, Marcickiewicz J, Gabel M, Groth K, Akouri R, Eklind S, Holgersson J, Tzakis A, Olausson M. First clinical uterus transplantation trial: a six-month report. Fertil Steril. 2014 May;101(5):1228-36. doi: 10.1016/j.fertnstert.2014.02.024. Epub 2014 Feb 27. PMID 24582522
- [Background] Ozturk H. How real is the uterine transplantation? Ann Transplant. 2014 Feb 14;19:82-3. doi: 10.12659/AOT.889973. No abstract available. PMID 24535028
- [Background] Akar ME, Ozkan O, Ozekinci M, Sindel M, Yildirim F, Oguz N. Uterus retrieval in cadaver: technical aspects. Clin Exp Obstet Gynecol. 2014;41(3):293-5. PMID 24992779
- [Derived] Fronek J, Janousek L, Kristek J, Chlupac J, Pluta M, Novotny R, Maluskova J, Olausson M. Live Birth Following Uterine Transplantation From a Nulliparous Deceased Donor. Transplantation. 2021 May 1;105(5):1077-1081. doi: 10.1097/TP.0000000000003346. PMID 32541565
- See also: Uterine transplantation in the Czech Republic, description and contacts — http://www.ikem.cz/en/transplantcentrum/klinika-transplantacni-chirurgie/o-nas/programy/transplantace-delohy/a-2460/